CLINICAL TRIAL: NCT06083987
Title: Optimizing Technology Interventions for Help-Seeking for Depression and Suicidality in Sexual and Gender Minority Youth
Brief Title: Sexual and Gender Minority Youth (SGMY) and Online Interventions to Increase Help-seeking for Anxiety and/or Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Ana Radovic, Assistant professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY22070134; 5R21MD015806-02 (NIH)
Record Dates: First submitted 2023-09-27; First posted 2023-10-16 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Depression; Adolescent Behavior; Sexual and Gender Minorities
MeSH Terms: conditions — Anxiety Disorders; Depression; Adolescent Behavior; Coitus | interventions — Confidentiality

STUDY DESIGN:
Intervention Model Description: 96 participants randomly assigned to one of the 16 combinations of the four study intervention principles
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Control Group - No Interventions (Active Comparator): Arm 1 will have not be given any of the interventions and will be a control group.
  Interventions: Behavioral: Control Group - No Interventions
- Intervention 1 - Intersectionality and Identity (Experimental): Arm 2 will be given access to intervention 1. It will have video and text content focused on identity and intersectionality.
  Interventions: Behavioral: Intersectionality and Identity
- Interventions 1 and 2 - Intersectionality and Identity/Confidentiality and Privacy (Experimental): Arm 3 will be given access to with the video and text content focused on intersectionality and confidentiality
  Interventions: Behavioral: Intersectionality and Identity; Behavioral: Confidentiality
- Interventions 1, 2, and 3 - Intersectionality/Confidentiality/Educational Tools (Experimental): Arm 4 will be given access to with the video and text content focused on intersectionality, confidentiality, and education about identity
  Interventions: Behavioral: Intersectionality and Identity; Behavioral: Confidentiality; Behavioral: Educating Your Community
- Interventions 1, 2, and 4 - Intersectionality/Confidentiality/Finding Affirming Care (Experimental): Arm 5 will be given access to interventions 1, 2, and 4, with the video and text content focused on intersectionality, confidentiality, and determining if caregivers are affirming
  Interventions: Behavioral: Intersectionality and Identity; Behavioral: Confidentiality; Behavioral: How to find Affirming Caregivers
- Interventions 1, 2, 3 and 4 - Intersectionality/Confidentiality/Educational Tools/Affirming Care (Experimental): Arm 6 will be given access to all 4 interventions, with the video and text content focused on intersectionality, confidentiality, education about identity, and determining if caregivers are affirming
  Interventions: Behavioral: Intersectionality and Identity; Behavioral: Confidentiality; Behavioral: Educating Your Community; Behavioral: How to find Affirming Caregivers
- Interventions 1 and 3 - Intersectionality and Identity/Educational Tools (Experimental): Arm 7 will be given access to interventions 1 and 3, with the video and text content focused on intersectionality and education about identity
  Interventions: Behavioral: Intersectionality and Identity; Behavioral: Educating Your Community
- Interventions 1, 3, and 4 - Intersectionality and Identity/Educational Tools/Finding Affirming Care (Experimental): Arm 8 will be given access to interventions 1, 3, and 4, with the video and text content focused on intersectionality, education about identity and determining if caregivers are affirming.
  Interventions: Behavioral: Intersectionality and Identity; Behavioral: Educating Your Community; Behavioral: How to find Affirming Caregivers
- Interventions 1 and 4 - Intersectionality and Identity/Finding Affirming Care (Experimental): Arm 9 will be given access to interventions 1 and 4, with the video and text content focused on intersectionality and determining if caregivers are affirming.
  Interventions: Behavioral: Intersectionality and Identity; Behavioral: How to find Affirming Caregivers
- Intervention 2 - Confidentiality and Privacy (Experimental): Arm 10 will be given access to intervention 2, with the video and text content focused on confidentiality
  Interventions: Behavioral: Confidentiality
- Interventions 2 and 3 - Confidentiality and Privacy/Educational Tools (Experimental): Arm 11 will be given access to interventions 2, and 3. Video and text content will focus on confidentiality and education about identity.
  Interventions: Behavioral: Confidentiality; Behavioral: Educating Your Community
- Interventions 2, 3 and 4 - Confidentiality and Privacy/Educational Tools/Finding Affirming Care (Experimental): Arm 12 will be given access to interventions 2, 3, and 4. Video and text content will focus on confidentiality, education about identity, and determine if caregivers are affirming.
  Interventions: Behavioral: Confidentiality; Behavioral: Educating Your Community; Behavioral: How to find Affirming Caregivers
- Interventions 2 and 4 - Confidentiality and Privacy/Finding Affirming Care (Experimental): Arm 13 will be given access to interventions 2 and 4. Video and text content will focus on confidentiality and determining if caregivers are affirming.
  Interventions: Behavioral: Confidentiality; Behavioral: How to find Affirming Caregivers
- Intervention 3 - Educational Tools (Experimental): Arm 14 will be given access to intervention 3. Video and text content will focus on education about identity
  Interventions: Behavioral: Educating Your Community
- Interventions 3 and 4 - Educational Tools/Finding Affirming Care (Experimental): Arm 15 will be given access to interventions 3 and 4. Video and text content will focus on educational tools about identity and determining if caregivers are affirming.
  Interventions: Behavioral: Educating Your Community; Behavioral: How to find Affirming Caregivers
- Intervention 4 - Finding Affirming Care (Experimental): Arm 16 will be given access to intervention 4, with video and text content focusing on determining if caregivers are affirming.
  Interventions: Behavioral: How to find Affirming Caregivers

INTERVENTIONS:
Behavioral: Intersectionality and Identity — Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of intersectionality and identity. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
  Arms: Intervention 1 - Intersectionality and Identity; Interventions 1 and 2 - Intersectionality and Identity/Confidentiality and Privacy; Interventions 1 and 3 - Intersectionality and Identity/Educational Tools; Interventions 1 and 4 - Intersectionality and Identity/Finding Affirming Care; Interventions 1, 2, 3 and 4 - Intersectionality/Confidentiality/Educational Tools/Affirming Care; Interventions 1, 2, and 3 - Intersectionality/Confidentiality/Educational Tools; Interventions 1, 2, and 4 - Intersectionality/Confidentiality/Finding Affirming Care; Interventions 1, 3, and 4 - Intersectionality and Identity/Educational Tools/Finding Affirming Care
Behavioral: Confidentiality — Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on Confidentiality for caregivers. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
  Arms: Intervention 2 - Confidentiality and Privacy; Interventions 1 and 2 - Intersectionality and Identity/Confidentiality and Privacy; Interventions 1, 2, 3 and 4 - Intersectionality/Confidentiality/Educational Tools/Affirming Care; Interventions 1, 2, and 3 - Intersectionality/Confidentiality/Educational Tools; Interventions 1, 2, and 4 - Intersectionality/Confidentiality/Finding Affirming Care; Interventions 2 and 3 - Confidentiality and Privacy/Educational Tools; Interventions 2 and 4 - Confidentiality and Privacy/Finding Affirming Care; Interventions 2, 3 and 4 - Confidentiality and Privacy/Educational Tools/Finding Affirming Care
Behavioral: Educating Your Community — Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of the education of family and friends about identity. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
  Arms: Intervention 3 - Educational Tools; Interventions 1 and 3 - Intersectionality and Identity/Educational Tools; Interventions 1, 2, 3 and 4 - Intersectionality/Confidentiality/Educational Tools/Affirming Care; Interventions 1, 2, and 3 - Intersectionality/Confidentiality/Educational Tools; Interventions 1, 3, and 4 - Intersectionality and Identity/Educational Tools/Finding Affirming Care; Interventions 2 and 3 - Confidentiality and Privacy/Educational Tools; Interventions 2, 3 and 4 - Confidentiality and Privacy/Educational Tools/Finding Affirming Care; Interventions 3 and 4 - Educational Tools/Finding Affirming Care
Behavioral: How to find Affirming Caregivers — Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of finding affirming caregivers. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
  Arms: Intervention 4 - Finding Affirming Care; Interventions 1 and 4 - Intersectionality and Identity/Finding Affirming Care; Interventions 1, 2, 3 and 4 - Intersectionality/Confidentiality/Educational Tools/Affirming Care; Interventions 1, 2, and 4 - Intersectionality/Confidentiality/Finding Affirming Care; Interventions 1, 3, and 4 - Intersectionality and Identity/Educational Tools/Finding Affirming Care; Interventions 2 and 4 - Confidentiality and Privacy/Finding Affirming Care; Interventions 2, 3 and 4 - Confidentiality and Privacy/Educational Tools/Finding Affirming Care; Interventions 3 and 4 - Educational Tools/Finding Affirming Care
Behavioral: Control Group - No Interventions — Control Group - Will be given no interventions
  Arms: Control Group - No Interventions

SUMMARY:
the investigators will use 4 technology based tools (combinations of youtube videos, links to online resources, tiktok videos, and other media) in a study of 96 Sexual and Gender Minority Youth (SGMY) to determine the effectiveness of them in helping youth to seek out mental health help. Participants will be divided into 1 of 16 groups and will interact with other participants anonymously on Discord. Each group will have access to 1, 2, 3, or all 4 of the tools which are categorized by a specific subject (except for one group who will have no access to the tools in order to compare this outcome against those who use the tools). There will be a survey before starting the Discord portion which will last 4 weeks, and a survey afterwards.

DETAILED DESCRIPTION:
Only one-third of adolescents access treatment for depression, and many fail to interact with clinic-based mental health resources. Sexual and gender minority youth (SGMY) are at greater risk for severe mental health disorders and suicidality but even less likely to access mental health services, even when access is available.

Widespread factors - stigma, negative beliefs about treatment, lack of mental health knowledge - contribute to not seeking services. Mainstream mental health interventions fail to address unique factors to SGMY that inhibit help-seeking: double stigma (stigma around mental health as well as internalized homophobia and transphobia), concern about revealing SGM status, low family support, lack of access to SGM affirming mental health professionals.

Despite being hard-to-reach, SGMY at risk for depression are quite active online. Yet SGMY-specific evidence-based online interventions are lacking and community interventions do not enhance mental health help-seeking. Targeted online interventions are needed to address unique factors which prevent help-seeking but are themselves usable and engaging. The current proposal will use a user-informed efficient approach to technology intervention design considering the heterogeneity and specific needs of SGMY. The investigators will use the Behavioral Intervention Technology Model to design and study several intervention principles (IPs), or theoretical concepts including intervention aims and behavioral strategies, to understand which mechanisms of action hold promise while being iterating design and potential modalities.

The investigators will use human computer interaction (HCI) framework, Discover, Design/Build, and Test to develop and study several IPs. Specifically, will use HCI techniques to develop initial prototypes and seek iterative user feedback and evaluate 4 finalized low-fidelity prototypes using a factorial trial to understand each IP prototype's individual and combined feasibility, usability, acceptability, and change in help-seeking intention in an online sample of diverse (racially, ethnically, age, gender identity, sexual orientation) SGMY.

This will inform the development of a high-fidelity intervention which may include different components for specific SGMY subgroups to be evaluated in a larger clinical trial. The PI, Dr. Radovic, is a physician researcher in adolescent medicine and has conducted years of research using stakeholder-informed methods and HCI techniques to inform intervention development. By working with experts in SGM health, stakeholder engagement, intervention design, qualitative analysis, HCI design, and BIT development and testing, the investigators have an exciting opportunity to bridge the gap for SGM adolescents with depression and suicidality to motivate and equip adolescents with the tools needed to access treatment.

This proposal is responsive to NOT-MH-18-031 by conducting nimble iterative testing and NOT-MD-19-001 - testing stigma reduction interventions. Adolescents who are sexual and gender minority (or LGBTQ) have rising rates of depression, anxiety, and suicidality but are less likely to get mental health treatment than other adolescents due to stigma and low family support. These adolescents are quite active online. This study aims to understand what types of technology interventions are most promising for helping them to seek mental health help when indicated.

Due to the exploratory nature of this clinical trial, we originally considered multiple secondary outcomes. As we proceeded with the study and obtained formative information from qualitative interviews to inform initial prototypes, we further clarified our conceptual model regarding our interests in the main outcome of mental health help-seeking and subsequent improvement in depression and anxiety symptoms. This help-seeking we hypothesized may be influenced by help-seeking intention, social support, internalized stigmatization of identity (internalized homophobia, internalized transphobia), confidentiality concerns, and expectations of rejection by mental healthcare providers. These measures therefore remained as secondary outcomes which we examined, and all others were moved to Other Pre-specified outcome measures.

With regards to statistical analysis, due to limitations in sample size, and non-normality of data, we used non-parametric tests of statistical significance within the primary outcome of mental health help-seeking intention between each intervention compared to not that intervention and adjusted for multiple tests using false-discovery rate q-value calculated with the Yekutieli method in Stata.

ELIGIBILITY:
List the inclusion criteria:

have access to a smartphone; have finished 6th grade; have access to and intellectual and physical ability to use the internet; fit demographic criteria (SGMY); and have symptoms of depression and/or anxiety that are mild or more severe (PHQ-8 and/or GAD-7 = 5 or above)

We will routinely monitor the sample to attempt to reach the following proportions:

50% ages 14-16 and 50% ages 17-19 50% identify as sexual minority but cisgender and 50% identify as not cisgender at least 40% identify as a racial or ethnic minority

If any of the proportions are reached (e.g. if 60% of recruited sample identify as not belonging to a racial or ethnic minority we will change screen settings to exclude those who are not

List the exclusion criteria:

no access to smart phone or internet, did not complete the 6th grade, not able to use internet, depression and anxiety are less than mild (PHQ-8 and GAD-7 scores <5); presently are in ongoing psychotherapy (i.e. have attended or plan to attend more than 1 session).

If they have been in therapy within the past 3 months

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Radovic, MD, MSc, Principal Investigator — University of Pittsburgh/UPMC
Locations (1):
- Virtual Social Media Based Recruitment, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Trial outcome data can be accessed by contacting the study principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon Completion of the study (estimated June 2024) and it will be available indefinitely via contacting Dr. Radovic
Access Criteria: Completed Data and results will be fully available upon request to any interested parties via email

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Attention Control Group: Arm 1 will only receive the control intervention.
  Individuals in the Attention Control Group will not be given any of the intervention content (1-4) and will receive video and text content focused on interest in research.
  Control group:
  Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of participating in research studies. Participants will receive one new video a week and will be asked to share their thoughts on research and past experiences with research.
- Arm 2: Intervention 1 - Intersectionality and Identity: Individuals in Arm 2 will receive Intervention 1 and will be exposed to video and text content focused on identity and intersectionality.
  Intersectionality and Identity: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of intersectionality and identity. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
- Arm 3: Intervention 1 + 2: Individuals in Arm 3 will receive both Intervention 1 (description in Arm 2 description box) and Intervention 2 (description in Arm 10 description box).
- Arm 4: Intervention 1 + 2 + 3: Individuals in Arm 4 will receive Intervention 1 (description in Arm 2 description box), Intervention 2 (description in Arm 10 description box) and Intervention 3 (description in Arm 14 description box).
- Arm 5: Intervention 1 + 2 + 4: Individuals in Arm 5 will receive Intervention 1 (description in Arm 2 description box), Intervention 2 (description in Arm 10 description box) and Intervention 4 (description in Arm 16 description box).
- Arm 6: Intervention 1 + 2 + 3 + 4: Individuals in Arm 6 will receive Intervention 1 (description in Arm 2 description box), Intervention 2 (description in Arm 10 description box) and Intervention 3 (description in Arm 14 description box) and Intervention 4 (description in Arm 16 description box).
- Arm 7: Intervention 1 + 3: Individuals in Arm 7 will receive Intervention 1 (description in Arm 2 description box), and Intervention 3 (description in Arm 14 description box).
- Arm 8: Intervention 1 + 3 + 4: Individuals in Arm 8 will receive Intervention 1 (description in Arm 2 description box), and Intervention 3 (description in Arm 14 description box) and Intervention 4 (description in Arm 16 description box).
- Arm 9: Intervention 1 + 4: Individuals in Arm 9 will receive Intervention 1 (description in Arm 2 description box), and Intervention 4 (description in Arm 16 description box).
- Arm 10: Intervention 2 - Confidentiality and Privacy: Arm 10 will be given access to intervention 2, with the video and text content focused on confidentiality
  Confidentiality: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on Confidentiality for caregivers. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
- Arm 11: Intervention 2 + 3: Individuals in Arm 11 will receive Intervention 2 (description in Arm 10 description box) and Intervention 3 (description in Arm 14 description box).
- Arm 12: Intervention 2 + 3 + 4: Individuals in Arm 12 will receive Intervention 2 (description in Arm 10 description box) and Intervention 3 (description in Arm 14 description box) and Intervention 4 (description in Arm 16 description box).
- Arm 13: Intervention 2 + 4: Individuals in Arm 13 will receive Intervention 2 (description in Arm 10 description box) and Intervention 4 (description in Arm 16 description box).
- Arm 14: Intervention 3 - Educational Tools: Arm 14 will be given access to intervention 3. Video and text content will focus on education about identity
  Educating Your Community: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of the education of family and friends about identity. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
- Arm 15: Intervention 3 + 4: Individuals in Arm 15 will receive Intervention 3 (description in Arm 14 description box) and Intervention 4 (description in Arm 16 description box).
- Arm 16: Intervention 4 - Finding Affirming Care: Arm 16 will be given access to intervention 4, with video and text content focusing on determining if caregivers are affirming.
  How to find Affirming Caregivers: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of finding affirming caregivers. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
Period: Overall Study
Arm/Group | Arm 1: Attention Control Group | Arm 2: Intervention 1 - Intersectionality and Identity | Arm 3: Intervention 1 + 2 | Arm 4: Intervention 1 + 2 + 3 | Arm 5: Intervention 1 + 2 + 4 | Arm 6: Intervention 1 + 2 + 3 + 4 | Arm 7: Intervention 1 + 3 | Arm 8: Intervention 1 + 3 + 4 | Arm 9: Intervention 1 + 4 | Arm 10: Intervention 2 - Confidentiality and Privacy | Arm 11: Intervention 2 + 3 | Arm 12: Intervention 2 + 3 + 4 | Arm 13: Intervention 2 + 4 | Arm 14: Intervention 3 - Educational Tools | Arm 15: Intervention 3 + 4 | Arm 16: Intervention 4 - Finding Affirming Care
Started | 4 | 5 | 5 | 5 | 5 | 6 | 6 | 5 | 4 | 6 | 5 | 4 | 5 | 5 | 6 | 5
Completed | 3 | 4 | 5 | 4 | 4 | 5 | 6 | 5 | 4 | 6 | 5 | 4 | 5 | 4 | 6 | 5
Not Completed | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Attention Control Group: Individuals in this group are individuals who are in Arm 1 and will only receive the control intervention.
  Individuals in the Attention Control Group will not be given any of the intervention content (1-4) and will receive video and text content focused on interest in research.
  Control group:
  Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of participating in research studies. Participants will receive one new video a week and will be asked to share their thoughts on research and past experiences with research.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Attention Control Group | Arm 2: Intervention 1 - Intersectionality and Identity | Arm 3: Intervention 1 + 2 | Arm 4: Intervention 1 + 2 + 3 | Arm 5: Intervention 1 + 2 + 4 | Arm 6: Intervention 1 + 2 + 3 + 4 | Arm 7: Intervention 1 + 3 | Arm 8: Intervention 1 + 3 + 4 | Arm 9: Intervention 1 + 4 | Arm 10: Intervention 2 - Confidentiality and Privacy | Arm 11: Intervention 2 + 3 | Arm 12: Intervention 2 + 3 + 4 | Arm 13: Intervention 2 + 4 | Arm 14: Intervention 3 - Educational Tools | Arm 15: Intervention 3 + 4 | Arm 16: Intervention 4 - Finding Affirming Care | Total
Number analyzed (Participants) | 4 | 5 | 5 | 5 | 5 | 6 | 6 | 5 | 4 | 6 | 5 | 4 | 5 | 5 | 6 | 5 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.3 (0.1) | 18.2 (1.3) | 17.6 (0.9) | 17.4 (1.3) | 18.2 (0.4) | 18.3 (0.5) | 18.5 (0.6) | 17.8 (1.3) | 18.2 (0.5) | 17.5 (0.8) | 18.4 (0.6) | 17.3 (2.2) | 18.2 (0.8) | 17.8 (1.1) | 18.3 (0.5) | 18.4 (0.9) | 18.0 (0.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 1 | 3 | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 2 | 3 | 1 | 2 | 24
  Male | 3 | 2 | 5 | 4 | 2 | 4 | 5 | 4 | 3 | 5 | 5 | 2 | 3 | 2 | 5 | 3 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 3 | 3 | 5 | 5 | 5 | 6 | 6 | 5 | 4 | 6 | 5 | 4 | 5 | 4 | 6 | 5 | 77
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 4 | 4 | 5 | 3 | 6 | 3 | 4 | 5 | 3 | 3 | 4 | 3 | 5 | 3 | 61
  White | 0 | 2 | 1 | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 15
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  Middle School (7-8th grade) | 0 | 0 | 3 | 0 | 2 | 2 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 2 | 1 | 16
  High School (9-12th grade) | 4 | 3 | 2 | 4 | 1 | 2 | 4 | 5 | 2 | 4 | 5 | 2 | 2 | 4 | 4 | 3 | 51
  Graduated High School | 0 | 2 | 0 | 1 | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 14
Easy Access to Transportation [Count of Participants; unit: Participants] | 4 | 3 | 5 | 5 | 4 | 6 | 6 | 5 | 4 | 6 | 5 | 4 | 4 | 5 | 5 | 4 | 75
MacArthur scale of subjective social status - United States [Mean (Standard Deviation); unit: units on a scale] — Asked to use a 1 to 10 ladder to rank one's social status as compared to everyone else in the United States; a higher rank indicates a higher social status; the range is 1-10
  units on a scale | 6 (0.7) | 6.0 (2.7) | 6.2 (0.4) | 6.2 (1.9) | 6.0 (0.7) | 6.0 (2.4) | 4.5 (1.5) | 4.2 (2.4) | 4.3 (1.5) | 6.3 (1.5) | 5.2 (1.6) | 5.3 (2.2) | 6.2 (1.3) | 5.0 (1.2) | 5.2 (1.3) | 5.4 (1.7) | 5.5 (0.2)
Ever Received Therapy [Count of Participants; unit: Participants] — ever receiving any psychotherapy
  Participants | 3 | 2 | 1 | 2 | 0 | 3 | 1 | 1 | 0 | 3 | 1 | 2 | 1 | 1 | 1 | 2 | 24
Ever Received Medication [Count of Participants; unit: Participants] — Ever receiving medication for a mental health concern
  Participants | 2 | 1 | 2 | 2 | 0 | 2 | 1 | 1 | 2 | 4 | 1 | 1 | 1 | 1 | 1 | 3 | 25
Access to Health Insurance [Count of Participants; unit: Participants] | 3 | 3 | 3 | 4 | 2 | 5 | 4 | 4 | 3 | 5 | 5 | 4 | 4 | 4 | 4 | 3 | 60
Have Primary Care Provider [Count of Participants; unit: Participants] | 4 | 4 | 4 | 4 | 3 | 6 | 6 | 4 | 3 | 6 | 5 | 4 | 4 | 4 | 5 | 4 | 70

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - IP Use Proportion
Description: Average proportions of IP components completed out of IP components available per individual participant (IP component defined as opportunity offered to interact with the intervention - some individuals will have more opportunities offered than others due to factorial randomization)
Time Frame: Over one month
Measure: Mean (Standard Deviation); unit: average proportion
Groups:
- Intervention 1: Individuals in this group receive Intervention 1 and will be exposed to video and text content focused on identity and intersectionality. They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
  Intervention 1 = Intersectionality and Identity: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of intersectionality and identity. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
- Intervention 2: Individuals in this group receive Intervention 2, with the video and text content focused on confidentiality.
  They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
  Intervention 2 = Confidentiality: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on Confidentiality for caregivers. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
- Intervention 3: Individuals in this group will receive Intervention 3. Video and text content will focus on education about identity. They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
  Intervention 3 = Educating Your Community: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of the education of family and friends about identity. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
- Intervention 4: Individuals in this group will receive Intervention 4, with video and text content focusing on determining if caregivers are affirming. They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
  Intervention 4 = How to find Affirming Caregivers: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of finding affirming caregivers. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
- Total Sample: Total Sample at Baseline
Arm/Group | Intervention 1 | Intervention 2 | Intervention 3 | Intervention 4 | Total Sample
Number analyzed (Participants) | 41 | 41 | 42 | 40 | 81
average proportion | 0.10 (0.17) | 0.11 (0.21) | 0.10 (0.16) | 0.08 (0.13) | 0.11 (0.19)

2. Primary Outcome: Feasibility - IP Use Days
Description: Average Proportion of days IP is used per individual (number of days session accessed over total offered which is 28 days)
Time Frame: Over one month
Population: Total sample who enrolled in the study; for this outcome all groups are combined because this was a feasibility metric of the entire pilot study population as a whole and not intended to compare across arms to answer the question, what proportion of days the study participants would access the online intervention?
Measure: Mean (Standard Deviation); unit: Mean proportion total days used per part
Arm/Group | Total Sample
Number analyzed (Participants) | 81
Mean proportion total days used per part | 0.04 (0.06)

3. Primary Outcome: Feasibility - IP Use Time
Description: Average length of time IP is used (length of session)
Time Frame: Over one month
Population: We do not have access to this data. Prior to starting the study, we had the understanding that we would be able to extract this level of data from the Discord platform. Upon beginning the study and collecting data, and after multiple iterative attempts, we were not able to obtain that data due to Discord regulations.
Groups:
- Full Sample: This is the full sample at baseline
Arm/Group | Full Sample
Number analyzed (Participants) | 0

4. Primary Outcome: Usability
Description: System Usability Scale, min: 0, Max: 100, higher scores mean better usability
Time Frame: 1 month
Population: For this outcome all groups are combined - for the full sample completing this follow-up measure. This was a usability metric of the entire pilot study population as a whole and not intended to compare across arms to answer the question, what is the usability rating of the entire online intervention?
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Full Sample Completing Follow-Up: This is the full sample completing this follow-up measure
Arm/Group | Full Sample Completing Follow-Up
Number analyzed (Participants) | 73
units on a scale | 77.4 (13.6)

5. Primary Outcome: Acceptability of the Intervention Principle
Description: Open-ended questions about whether the Discord server and the tools used were: helpful; whether it was affirming of SGM status; if timing and amount of content were appropriate, if privacy and confidentiality were maintained, and if they had any negative consequences of participation (e.g. parent questioning them )
Time Frame: 1 month
Population: For this outcome all groups are combined - for the full sample completing this follow-up measure. This was acceptability metric was of the entire pilot study population as a whole and not intended to compare across arms to answer the question, what is the acceptability rating of the entire online intervention?
Measure: Count of Participants; unit: Participants
Arm/Group | Full Sample Completing Follow-Up
Number analyzed (Participants) | 75
Participants
  Felt Discord Server and Tools were Helpful | 72
  Felt Content was Appropriate | 74
  Timing of Posting/Receiving Content Appropriate | 73
  Felt Affirmed (received emotional support or encouragement) about your sexuality or gender | 73
  Felt Privacy and Confidentiality were Maintained | 74
  Experienced any Negative Consequences from Participation | 0

6. Primary Outcome: Help-Seeking Intention From Counselor or Therapist - TAU vs Not TAU
Description: single help-seeking intention ruler-based question (i.e. 'I intend to seek help from a counselor or therapist for my mental health problems' scale 1-7, a higher number signifying a higher intent to seek help
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment as Usual (TAU): Individuals in this group only completed treatment as usual (did not receive any Intervention 1 through 4 but just participated in the Discord Server research channel. Also completed follow up measures.
- Not TAU (Treatment As Usual): Individuals in this group include all other participants who did not receive treatment as usual only and completed follow up measures
Arm/Group | Treatment as Usual (TAU) | Not TAU (Treatment As Usual)
Number analyzed (Participants) | 3 | 72
units on a scale | 4.00 (1.00) | 3.99 (1.30)
Statistical Analysis 1: Comparison: Treatment as Usual (TAU) vs Not TAU (Treatment As Usual); Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney); false discovery rate q-value calculated with Yekutieli method in Stata; Cohen's D = 0.01

7. Primary Outcome: Help-Seeking Intention From Counselor or Therapist - Intervention 1 vs. Not 1
Description: as for outcome 6
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention 1: Individuals in this group receive Intervention 1 and completed follow up measures. They were exposed to video and text content focused on identity and intersectionality. They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
  Intervention 1 = Intersectionality and Identity: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of intersectionality and identity. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
- Not Intervention 1: Individuals in this group include all other participants who did not receive intervention 1 but completed follow up measures
Arm/Group | Intervention 1 | Not Intervention 1
Number analyzed (Participants) | 37 | 38
units on a scale | 4.19 (1.19) | 3.79 (1.36)
Statistical Analysis 1: Comparison: Intervention 1 vs Not Intervention 1; Test type: Superiority; p = 0.31, Wilcoxon (Mann-Whitney); Cohen's D = 0.32

8. Primary Outcome: Help-Seeking Intention From Counselor or Therapist - Intervention 2 vs. Not 2
Description: as for outcome 6
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention 2: Individuals in this group receive Intervention 2 and completed follow up measures.
  Individuals in this group receive Intervention 2, with the video and text content focused on confidentiality.
  They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
  Intervention 2 = Confidentiality: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on Confidentiality for caregivers. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
- Not Intervention 2: Individuals in this group include all other participants who did not receive intervention 2 but completed follow up measures
Arm/Group | Intervention 2 | Not Intervention 2
Number analyzed (Participants) | 38 | 37
units on a scale | 4.05 (1.37) | 3.92 (1.21)
Statistical Analysis 1: Comparison: Intervention 2 vs Not Intervention 2; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney); Cohen's D = 0.10

9. Primary Outcome: Help-Seeking Intention From Counselor or Therapist - Intervention 3 vs. Non-3
Description: as for outcome 6
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention 3: Individuals in this group receive Intervention 3 and completed follow up measures.
  Individuals in this group will receive Intervention 3. Video and text content will focus on education about identity. They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
  Intervention 3 = Educating Your Community: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of the education of family and friends about identity. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
- Not Intervention 3: Individuals in this group include all other participants who did not receive intervention 3 but completed follow up measures
Arm/Group | Intervention 3 | Not Intervention 3
Number analyzed (Participants) | 39 | 36
units on a scale | 4.26 (1.14) | 3.69 (1.39)
Statistical Analysis 1: Comparison: Intervention 3 vs Not Intervention 3; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney); Cohen's D = 0.45

10. Primary Outcome: Help-Seeking Intention From Counselor or Therapist - Intervention 4 vs. Not 4
Description: as for outcome 6
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention 4: Individuals in this group receive Intervention 4 and completed follow up measures.
  Individuals in this group will receive Intervention 4, with video and text content focusing on determining if caregivers are affirming. They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
  Intervention 4 = How to find Affirming Caregivers: Participants will use the computer application, Discord, a social media site that allows for sharing of content and interaction with other people in a variety of forms (video chat, direct messaging, and talking in group chat areas). We will be using the group chat function to set up discussion forums where there will be video and text resources focused on matters of finding affirming caregivers. Participants will do at least one activity from three types each week for four weeks. The three activity types will have the participants engage with the content and then either discuss it in the forum ("Talk about it"), write a review about the content discussing why/why not they like it ("Rate it"), or Attempt to use the knowledge or skills to accomplish a task offline ("Try it").
- Not Intervention 4: Individuals in this group include all other participants who did not receive intervention 4 but completed follow up measures
Arm/Group | Intervention 4 | Not Intervention 4
Number analyzed (Participants) | 38 | 37
units on a scale | 4.24 (1.05) | 3.72 (1.47)
Statistical Analysis 1: Comparison: Intervention 4 vs Not Intervention 4; Test type: Superiority; p = 0.22, Wilcoxon (Mann-Whitney); Cohen's d = 0.41

11. Secondary Outcome: Social Support - TAU vs Not TAU
Description: The Medical Outcome Study Social Support Scale measures types of social support. Per item, options range from 1 to 5 with higher levels are associated with greater support. We will use the emotional/informational subscale from this report and instead of transforming to 0-100 like the original, we will use the untransformed mean score of the items which can range 1 to 5.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual (TAU) | Not TAU (Treatment As Usual)
Number analyzed (Participants) | 3 | 72
units on a scale | 3.54 (1.08) | 3.45 (0.78)

12. Secondary Outcome: Social Support - Intervention 1 vs. Not 1
Description: as for outcome 11
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention 1 | Not Intervention 1
Number analyzed (Participants) | 37 | 38
units on a scale | 3.57 (0.78) | 3.35 (0.78)

13. Secondary Outcome: Social Support - Intervention 2 vs. Not 2
Description: as for outcome 11
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention 2: Individuals in this group receive Intervention 2 and completed follow up measures.
  Individuals in this group receive Intervention 2, with the video and text content focused on confidentiality.
  They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
Arm/Group | Intervention 2 | Not Intervention 2
Number analyzed (Participants) | 38 | 37
units on a scale | 3.41 (0.78) | 3.51 (0.79)

14. Secondary Outcome: Social Support - Intervention 3 vs. Not 3
Description: as for outcome 11
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention 3: Individuals in this group receive Intervention 3 and completed follow up measures.
  Individuals in this group will receive Intervention 3. Video and text content will focus on education about identity. They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
Arm/Group | Intervention 3 | Not Intervention 3
Number analyzed (Participants) | 39 | 36
units on a scale | 3.38 (0.77) | 3.53 (0.79)

15. Secondary Outcome: Social Support - Intervention 4 vs. Not 4
Description: as for outcome 11
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention 4: Individuals in this group receive Intervention 4 and completed follow up measures.
  Individuals in this group will receive Intervention 4, with video and text content focusing on determining if caregivers are affirming. They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
Arm/Group | Intervention 4 | Not Intervention 4
Number analyzed (Participants) | 38 | 37
units on a scale | 3.61 (0.82) | 3.30 (0.72)

16. Secondary Outcome: Internalized Homophobia - TAU vs Not TAU
Description: Sexual Minority Adolescent Stress Inventory Internalized homonegativity subscale for the past 30 days. min: 0, max: 7. Higher score indicates greater internalized homophobia
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) | Not TAU (Treatment As Usual)
Number analyzed (Participants) | 3 | 72
score on a scale | 1.00 (1.73) | 0.69 (0.99)

17. Secondary Outcome: Internalized Homophobia - Intervention 1 vs Not 1
Description: Sexual Minority Adolescent Stress Inventory Internalized homonegativity subscale. - asked about past 30 days min: 0, max: 7. Higher score indicates greater internalized homophobia
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention 1: Individuals in this group receive Intervention 1 and completed follow up measures. They were exposed to video and text content focused on identity and intersectionality. They may or may not receive additional interventions. These groups will overlap due to the factorial design and some individuals receiving more than one Intervention.
Arm/Group | Intervention 1 | Not Intervention 1
Number analyzed (Participants) | 37 | 38
score on a scale | 0.68 (0.97) | 0.74 (1.06)

18. Secondary Outcome: Internalized Homophobia - Intervention 2 vs Not 2
Description: as for outcome 17
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 2 | Not Intervention 2
Number analyzed (Participants) | 38 | 37
score on a scale | 0.76 (1.00) | 0.65 (1.03)

19. Secondary Outcome: Internalized Homophobia - Intervention 3 vs Not 3
Description: as for outcome 17
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 3 | Not Intervention 3
Number analyzed (Participants) | 39 | 36
score on a scale | 0.77 (1.09) | 0.64 (0.93)

20. Secondary Outcome: Internalized Homophobia - Intervention 4 vs Not 4
Description: as for outcome 17
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 4 | Not Intervention 4
Number analyzed (Participants) | 38 | 37
score on a scale | 0.68 (0.93) | 0.73 (1.10)

21. Secondary Outcome: Internalized Transphobia - TAU vs Not TAU
Description: Gender Minority Stress and Resilience Measure. min: 0, max: 40. Higher score indicates greater internalized transphobia
Time Frame: 1 month
Population: this is the population which identified as transgender/nonbinary/gender-diverse
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) | Not TAU (Treatment As Usual)
Number analyzed (Participants) | 2 | 36
score on a scale | 7.00 (1.41) | 9.53 (7.92)

22. Secondary Outcome: Internalized Transphobia - Intervention 1 vs Not 1
Description: Gender Minority Stress and Resilience Measure. min: 0, max: 40. Higher score indicates greater internalized transphobia
Time Frame: 1 month
Population: this is the population which identified as transgender/nonbinary/gender-diverse
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 1 | Not Intervention 1
Number analyzed (Participants) | 17 | 21
score on a scale | 7.59 (5.78) | 10.86 (8.88)

23. Secondary Outcome: Internalized Transphobia - Intervention 2 vs Not 2
Description: Gender Minority Stress and Resilience Measure. min: 0, max: 40. Higher score indicates greater internalized transphobia
Time Frame: 1 month
Population: this is the population which identified as transgender/nonbinary/gender-diverse
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 2 | Not Intervention 2
Number analyzed (Participants) | 21 | 17
score on a scale | 10.62 (7.94) | 7.88 (7.42)

24. Secondary Outcome: Internalized Transphobia - Intervention 3 vs Not 3
Description: Gender Minority Stress and Resilience Measure. min: 0, max: 40. Higher score indicates greater internalized transphobia
Time Frame: 1 month
Population: this is the population which identified as transgender/nonbinary/gender-diverse
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Not Intervention 3: Not Intervention 3 Individuals in this group include all other participants who did not receive intervention 3 but completed follow up measures
Arm/Group | Intervention 3 | Not Intervention 3
Number analyzed (Participants) | 15 | 23
score on a scale | 11.8 (9.72) | 7.83 (5.82)

25. Secondary Outcome: Internalized Transphobia - Intervention 4 vs Not 4
Description: Gender Minority Stress and Resilience Measure. min: 0, max: 40. Higher score indicates greater internalized transphobia
Time Frame: 1 month
Population: this is the population which identified as transgender/nonbinary/gender-diverse
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 4 | Not Intervention 4
Number analyzed (Participants) | 18 | 20
score on a scale | 8.89 (8.51) | 9.85 (7.15)

26. Secondary Outcome: Expectance of Rejection Due to SGM Status TAU vs Not TAU
Description: Single-item yes/no and open ended question - asked about past 30 days
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual (TAU) | Not TAU (Treatment As Usual)
Number analyzed (Participants) | 3 | 72
Participants | 1 | 17

27. Secondary Outcome: Expectance of Rejection Due to SGM Status Intervention 1 vs Not 1
Description: Single-item yes/no and open ended question - asked about past 30 days
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention 1 | Not Intervention 1
Number analyzed (Participants) | 37 | 38
Participants | 8 | 10

28. Secondary Outcome: Expectance of Rejection Due to SGM Status Intervention 2 vs Not 2
Description: Single-item yes/no and open ended question - asked about past 30 days
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention 2 | Not Intervention 2
Number analyzed (Participants) | 38 | 37
Participants | 9 | 9

29. Secondary Outcome: Expectance of Rejection Due to SGM Status Intervention 3 vs Not 3
Description: Single-item yes/no and open ended question - asked about past 30 days
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention 3 | Not Intervention 3
Number analyzed (Participants) | 39 | 36
Participants | 10 | 8

30. Secondary Outcome: Expectance of Rejection Due to SGM Status Intervention 4 vs Not 4
Description: Single-item yes/no and open ended question - asked about past 30 days
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention 4 | Not Intervention 4
Number analyzed (Participants) | 38 | 37
Participants | 9 | 9

31. Secondary Outcome: Confidentiality Concerns TAU vs Not TAU
Description: Confidentiality item from BASH-B scale, min: 1, max: 6, higher score means individual agrees that a therapist would not maintain confidentiality
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual (TAU) | Not TAU (Treatment As Usual)
Number analyzed (Participants) | 3 | 72
units on a scale | 3 (1) | 2.53 (1.16)

32. Secondary Outcome: Confidentiality Concerns Intervention 1 vs Not 1
Description: as for outcome 31
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention 1 | Not Intervention 1
Number analyzed (Participants) | 37 | 38
units on a scale | 2.43 (1.24) | 2.66 (1.07)

33. Secondary Outcome: Confidentiality Concerns Intervention 2 vs Not 2
Description: as for outcome 31
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention 2 | Not Intervention 2
Number analyzed (Participants) | 38 | 37
units on a scale | 2.42 (1.15) | 2.68 (1.16)

34. Secondary Outcome: Confidentiality Concerns Intervention 3 vs Not 3
Description: as for outcome 31
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention 3 | Not Intervention 3
Number analyzed (Participants) | 39 | 36
units on a scale | 2.59 (1.23) | 2.50 (1.08)

35. Secondary Outcome: Confidentiality Concerns Intervention 4 vs Not 4
Description: as for outcome 31
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention 4 | Not Intervention 4
Number analyzed (Participants) | 38 | 37
units on a scale | 2.50 (1.16) | 2.59 (1.17)

36. Secondary Outcome: Receipt of Any Mental Health Treatment in Past 4 Weeks TAU vs Not TAU
Description: Actual Help Seeking Questionnaire (Rickwood 2005) which does not involve scoring; list of whether help-seeking was sought from different individuals for mental health concerns
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual (TAU) | Not TAU (Treatment As Usual)
Number analyzed (Participants) | 3 | 72
Participants | 1 | 30

37. Secondary Outcome: Receipt of Any Mental Health Treatment in Past 4 Weeks Intervention 1 vs Not 1
Description: as for outcome 36
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention 1 | Not Intervention 1
Number analyzed (Participants) | 37 | 38
Participants | 15 | 16

38. Secondary Outcome: Receipt of Any Mental Health Treatment in Past 4 Weeks Intervention 2 vs Not 2
Description: as for outcome 36
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention 2 | Not Intervention 2
Number analyzed (Participants) | 38 | 37
Participants | 16 | 15

39. Secondary Outcome: Receipt of Any Mental Health Treatment in Past 4 Weeks Intervention 3 vs Not 3
Description: as for outcome 36
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention 3 | Not Intervention 3
Number analyzed (Participants) | 39 | 36
Participants | 18 | 13

40. Secondary Outcome: Receipt of Any Mental Health Treatment in Past 4 Weeks Intervention 4 vs Not 4
Description: as for outcome 36
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention 4 | Not Intervention 4
Number analyzed (Participants) | 38 | 37
Participants | 16 | 15

41. Secondary Outcome: Depression Symptoms TAU vs Not TAU
Description: Patient Health Questionnaire-8 measures depression severity with a score ranging from 0 to 24, a higher score indicating greater severity.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) | Not TAU (Treatment As Usual)
Number analyzed (Participants) | 3 | 72
score on a scale | 4.33 (3.51) | 6.01 (4.22)

42. Secondary Outcome: Depression Symptoms Intervention 1 vs Not 1
Description: as for outcome 41
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 1 | Not Intervention 1
Number analyzed (Participants) | 37 | 38
score on a scale | 5.76 (4.03) | 6.13 (4.39)

43. Secondary Outcome: Depression Symptoms Intervention 2 vs Not 2
Description: as for outcome 41
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 2 | Not Intervention 2
Number analyzed (Participants) | 38 | 37
score on a scale | 6.13 (4.69) | 5.76 (3.66)

44. Secondary Outcome: Depression Symptoms Intervention 3 vs Not 3
Description: as for outcome 41
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 3 | Not Intervention 3
Number analyzed (Participants) | 39 | 36
score on a scale | 5.38 (3.51) | 6.56 (4.8)

45. Secondary Outcome: Depression Symptoms Intervention 4 vs Not 4
Description: as for outcome 41
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 4 | Not Intervention 4
Number analyzed (Participants) | 38 | 37
score on a scale | 6.00 (4.12) | 5.89 (4.32)

46. Secondary Outcome: Anxiety Symptoms - TAU vs Not TAU
Description: Generalized Anxiety Disorders 7-item Questionnaire measures extent of anxiety symptoms. The total score ranges from 0 to 21 with a higher score indicating greater severity.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment as Usual (TAU) | Not TAU (Treatment As Usual)
Number analyzed (Participants) | 3 | 72
score on a scale | 4.67 (3.21) | 5.23 (3.81)

47. Other Pre Specified Outcome: Social Isolation
Description: 4-item version of revised UCLA Loneliness Scale. min: 4, max: 16. Higher score means greater levels of loneliness
Time Frame: 1 month
Reporting Status: Not Posted

48. Other Pre Specified Outcome: Antidepressant Outcome Expectations
Description: The Antidepressant Meanings Scale (Cohane, 2008) measures an individual's level of negative attitudes toward taking an antidepressant medication if prescribed. It is a continuous measure and the total score ranges from 0 to 24, with a higher score indicating more negative attitudes.
Time Frame: 1 month
Reporting Status: Not Posted

49. Other Pre Specified Outcome: Beliefs About Therapy
Description: Barriers to Adolescents Seeking Help Scale-Brief Version (Wilson 2005/Kuhl 1997) measures perceptions about seeking treatment from a mental health provider. The total score ranges from 1 to 11, a higher score indicated greater barriers.
Time Frame: 1 month
Reporting Status: Not Posted

50. Other Pre Specified Outcome: 12 Item Short Form Survey From the RAND Medical Outcomes Study (SF-12)
Description: SF-12 (Jenkinson 1997).
  SF-12 survey generates two summary scores: a physical component score (pcs-12) and a mental component score (mcs-12). These scores are calculated using an algorithm that weighs the responses according to their contribution to the physical or mental health dimensions. The scores are then standardized to have a mean of 50 and a standard deviation of 10 in the general population. Higher scores indicate better health status and lower scores worse health status.
  PCS-12 raw scores min is -3.37 and max is 69.68.
  MCS-12 raw scores min is -10.64 and max is 73.18
Time Frame: 1 month
Reporting Status: Not Posted

51. Other Pre Specified Outcome: Mental Health Stigma, Personal and Perceived
Description: The Depression Stigma Scale (Griffiths 2004) measures stigmatizing attitudes toward depression treatment. It is a continuous measure and the total score ranges from 0-36. There are two subscales: the personal stigma subscale which totals 0-18 and the perceived stigma subscale which totals 0-18. These two are summed for the total stigma score. A higher score indicates a worse outcome.
Time Frame: 1 month
Reporting Status: Not Posted

52. Other Pre Specified Outcome: Perceived Need for Treatment
Description: Open-ended question about whether adolescent thinks they need any mental health service
Time Frame: 1 month
Reporting Status: Not Posted

53. Other Pre Specified Outcome: Help-Seeking Intention From Multiple Sources
Description: The General Help Seeking Questionnaire (Rickwood, 2005) asks the likelihood of seeking help from a potential individual for a personal or emotional problem. A higher score per individual indicates a higher likelihood and intention to seek help from this source.
Time Frame: 1 month
Reporting Status: Not Posted

54. Other Pre Specified Outcome: Depression and Anxiety Knowledge
Description: The Depression and Anxiety literacy questionnaires (Gulliver 2012) measures knowledge about depression and anxiety diagnosis and treatment. The total score ranges from 0-22, with a higher score indicating greater knowledge of depression. We will use a brief version of this scale.
Time Frame: 1 month
Reporting Status: Not Posted

55. Secondary Outcome: Anxiety Symptoms - Intervention 1 vs Not 1
Description: as for outcome 46
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 1 | Not Intervention 1
Number analyzed (Participants) | 37 | 38
score on a scale | 4.95 (3.74) | 5.65 (3.82)

56. Secondary Outcome: Anxiety Symptoms - Intervention 2 vs Not 2
Description: as for outcome 46
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 2 | Not Intervention 2
Number analyzed (Participants) | 38 | 37
score on a scale | 5.63 (4.46) | 4.94 (2.91)

57. Secondary Outcome: Anxiety Symptoms - Intervention 3 vs Not 3
Description: as for outcome 46
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 3 | Not Intervention 3
Number analyzed (Participants) | 39 | 36
score on a scale | 4.97 (3.66) | 5.64 (3.91)

58. Secondary Outcome: Anxiety Symptoms - Intervention 4 vs Not 4
Description: as for outcome 46
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention 4 | Not Intervention 4
Number analyzed (Participants) | 38 | 37
score on a scale | 5.00 (3.81) | 5.61 (3.77)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Full Sample: This is the full sample at baseline. Groups are not described separately because adverse outcomes for this pilot trial were not expected to differ based on study arm and so therefore adverse event data were collected irrespective of study arm - as only content per arm varied but everyone was exposed to the same intervention structure.
Arm/Group | Full Sample
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT06083987/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT06083987/ICF_002.pdf